CLINICAL TRIAL: NCT01598142
Title: Single-operator Wire-guided ERCP Cannulation Technique: a Single-center Randomized Controlled Study
Brief Title: Single-operator Wire-guided Endoscopic Retrograde Cholangiopancreatography Cannulation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qi-yong Li (Other)
Responsible Party: Sponsor-Investigator, Qi-yong Li, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YLS2011-105
Record Dates: First submitted 2011-11-01; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Biliary Diseases; Pancreas Diseases
Keywords: Endoscopic retrograde cholangiopancreatography (ERCP); Guidewires; Cannulation; Single-operator; C-Hook
MeSH Terms: conditions — Gallbladder Diseases; Pancreatic Diseases | interventions — Coping Orientation to Problems Experienced Questionnaire

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experienced assistant group (Other): experienced endoscopist with an experienced assistant.
  Interventions: Procedure: Team 1
- new trained assistant group (Other): same experienced endoscopist with a new trained assistant
  Interventions: Procedure: Team 2

INTERVENTIONS:
Procedure: Team 1 — experienced endoscopist with a experienced assistant
  Other Names: experienced
  Arms: experienced assistant group
Procedure: Team 2 — same experienced endoscopist with a new trained assistant
  Other Names: new trained
  Arms: new trained assistant group

SUMMARY:
The single-operator wire-guided cannulation technique doesn't require an experienced assistant and precise coordination between the assistant and endoscopist.

DETAILED DESCRIPTION:
A new single-operator wire-guided cannulation technique was performed on all patients. All procedures were performed by the same experienced endoscopist, but with different assistants in two groups (with an experienced one in Group A, and a new trained one in Group B). The number of attempts at cannulation, cannulation time, success rate, and procedure-related complications were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with pancreas and biliary diseases referred to the authors for ERCP

Exclusion Criteria:

* previous endoscopic sphincterotomy,
* surgically altered anatomy (e.g. Billroth II gastrectomy) or
* diagnostic duodenoscopy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Cannulation success rate | two years

SECONDARY OUTCOMES:
Incidences of post-ERCP pancreatitis | two years
Incidences of bleeding | two years
Incidences of perforation | two years
Incidences of infection | two years
Number of attempts at cannulation | two years
Cannulation time | two years

CONTACTS AND LOCATIONS:
Overall Officials: Qi-Yong Li, MD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China